CLINICAL TRIAL: NCT01643616
Title: Ultrasound Guided Distal Sciatic Nerve Block - a Randomised Comparison With Nerve Stimulator Technique
Brief Title: Ultrasound Guided Distal Sciatic Nerve Block - a Comparison With Nerve Stimulator Technique
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Research Center (Other)
Responsible Party: Principal Investigator, Dr.med.Ronald Seidel, Dr.med.Ronald Seidel, Helios Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HV 2010 003
Record Dates: First submitted 2012-07-16; First posted 2012-07-18 (Estimated); Results first posted 2013-11-01 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-08

CONDITIONS: Other Surgical Procedures
Keywords: Sciatic Nerve; Ultrasound; Anesthesia, Regional; Orthopedic Surgery
MeSH Terms: interventions — Midazolam; Prilocaine; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- group US (Active Comparator): Ultrasound guided block :
  20ml Prilocaine 1% and 10ml Ropivacaine 0.75% (30ml Prilocaine 1% in outpatients)
  Interventions: Drug: midazolam; Drug: Prilocaine 1%; Drug: Ropivacaine 0.75%; Device: ultrasound guidance
- group NS (Active Comparator): Nerve stimulation technique:
  20ml Prilocaine 1% and 10ml Ropivacaine 0.75% (30ml Prilocaine 1% in outpatients)
  Interventions: Drug: midazolam; Drug: Prilocaine 1%; Drug: Ropivacaine 0.75%; Device: nerve stimulation technique

INTERVENTIONS:
Drug: midazolam — Prior to performing the regional anesthesia the investigators administered midazolam as a premedication by mouth (3,75-7,5mg) or intravenously (2-3mg).
  Other Names: Dormicum
Drug: Prilocaine 1% — 20ml Prilocaine 1% for distal sciatic nerve block (30ml Prilocaine 1% in outpatients)
  Other Names: Xylonest
Drug: Ropivacaine 0.75% — 10ml Ropivacaine 0.75% for distal sciatic nerve block (not in outpatients)
  Other Names: Naropin
Drug: Prilocaine 1% — 10ml Prilocaine 1% for saphenous nerve block
  Other Names: Xylonest
Device: ultrasound guidance — In group US the sciatic nerve localization and needle guidance is realized using ultrasound.
  Arms: group US
Device: nerve stimulation technique — In the group NS sciatic nerve localization and needle guidance is realized using nerve stimulation technique. However, ultrasound is used observing (Observer) the procedure, but blinded for the physician (Anesthetist) performing the block.
  Arms: group NS

SUMMARY:
For distal sciatic nerve block this prospective, randomised comparison with ultrasound guided distal subepineural block tested the hypothesis, that intraepineural injection of local anesthetic using nerve stimulation technique is common and associated with high success rate.

DETAILED DESCRIPTION:
Classical methods for nerve localization (loss of resistance, cause of paresthesias, nerve stimulation technique)assumed that the target is a close approximation to the nerve, without epineural perforation. Intraneural injections were considered as evitable, with high risk for nerve damages.

Ultrasound guidance provided for the first time a real-time visualization of the spread of local anesthetic. Some recent studies proved, that an intraneural injection using nerve stimulator technique is common and not necessarily accompanied with nerve damages.

In the ultrasound group (group US) the investigators tested the hypothesis, that an intraneural injection of local anesthetic generate a high success rate and a short onset time without clinical apparent nerve damages.

In the nerve-stimulation group (group NS) the investigators tested the hypothesis, that an intraneural injection of local anesthetic is common, and in case of intraneural injection accompanied likewise with high success rate and shorter onset time.

For the sciatic division the investigators tested the hypothesis, that classical methods of nerve localization (nerve-stimulation technique, cause of paresthesias) are not able to avoid epineural perforation.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery on the foot or ankle
* tourniquet distal of the knee
* adult patients, 18-75 years old
* ASA-risk-groups I-III (American Society of Anesthesiologists)
* informed consent

Exclusion Criteria:

* severe coagulopathy
* systemic inflammatory response
* ASA-risk-groups > III (American Society of Anesthesiologists)
* drug allergy: local anesthetics
* pregnancy, lactation period
* participation in other studies
* addiction to drugs or alcohol
* non-cooperative patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2010-11; Primary Completion 2012-06 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Seidel, Dr. med., Principal Investigator — Klinik für Anästhesiologie und Intensivtherapie, Helios Kliniken Schwerin, Wismarsche Strasse 393-7, DE-19049 Schwerin; Georg Rehmert, Dr. med., Study Director — Klinik für Anästhesiologie und Intensivtherapie, Helios Kliniken Schwerin, Wismarsche Strasse 393-7, DE-19049 Schwerin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients were informed and included in the study in the anesthesiology outpatient clinic as part of normal pre-operative preparation. Using a computer-generated list of random numbers, patients were randomly allocated to either the nerve stimulation group (NS group, n=125) or the ultrasound group (US group, n=125).
Period: Overall Study
Arm/Group | Group US | Group NS
Started | 125 | 125
Completed | 125 | 125
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group US | Group NS | Total
Number analyzed (Participants) | 125 | 125 | 250
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 99 | 95 | 194
  >=65 years | 26 | 30 | 56
Age Continuous [Mean (Standard Deviation); unit: years] | 53.4 (14.3) | 56.4 (11.8) | 54.9 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 91 | 198
  Male | 18 | 34 | 52
Region of Enrollment [Number; unit: participants]
  Germany | 125 | 125 | 250

OUTCOME MEASURES:

1. Primary Outcome: Success Rate Without Supplementation
Description: After injection of local anesthetic a waiting period of 30-60 minutes was defined before completing a failed block.
  1. success without supplementation = no additional analgetics or rescue blocks required (success rate without supplementation, outcome measure 1)
  2. success with supplementation = analgetics or selective rescue blocks distal of the sciatic division required (success rate without supplementation and additionally all supplemented blocks, outcome measure 3)
  3. failed block = change of anesthetic procedure (general, spinal) or rescue blocks proximal of the sciatic division
Time Frame: within 30-60 minutes after injection of the local anesthetic
Population: In the NS group two investigators were necessary in order to realize the blinded study protocol. For personnel reasons this was not possible in every case and led to deviations from the randomization protocol for seven patients in each group. These patients were excluded from the analysis.
Measure: Number; unit: participants
Arm/Group | Group US | Group NS
Number analyzed (Participants) | 118 | 118
participants | 112 | 73
Statistical Analysis 1: Comparison: Group US vs Group NS; For sample size calculation we assumed a significance level of 0.05 and a success rate derived from clinical data of 75% in the nerve stimulation group and of 90% in the ultrasound group. With a group ratio of 1:1 and a power of 0.8, the required sample size was at least 226. For statistical analysis we used the exact Fisher test as a distribution-free, non-parametric test method; Test type: Superiority or Other; p < 0.05, Fisher Exact; Percentage Difference = 33 — For success rate without supplementation the difference between group US (94.9%) and group NS (61.9%) is 33%

2. Primary Outcome: Time Until Readiness for Surgery (Minutes)
Time Frame: within 60 minutes after injection of the local anesthetic
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Group US | Group NS
Number analyzed (Participants) | 118 | 118
minutes | 15.1 [13.6 to 16.5] | 28 [24.9 to 31.1]
Statistical Analysis 1: Comparison: Group US vs Group NS; We used the log-rank test to compare the onset times. The significance level was defined with p<0.05; Test type: Superiority or Other; p < 0.05, Log Rank; Mean Difference (Final Values) = 22.9, 95% CI 2-sided [13.6 to 31.1]

3. Primary Outcome: Success Rate With Supplementation
Description: After injection of local anesthetic a waiting period of 30-60 minutes was defined before completing a failed block.
  1. success without supplementation = no additional analgetics or rescue blocks required (success rate without supplementation, outcome measure 1)
  2. success with supplementation = analgetics or selective rescue blocks distal of the sciatic division required (success rate without supplementation and additionally all supplemented blocks, outcome measure 3)
  3. failed block = change of anesthetic procedure (general, spinal) or rescue blocks proximal of the sciatic divisionSucces rate with supplementation
Time Frame: later than 30-60 minutes after injection of the local anesthetic
Measure: Number; unit: participants
Arm/Group | Group US | Group NS
Number analyzed (Participants) | 118 | 118
participants | 116 | 85
Statistical Analysis 1: Comparison: Group US vs Group NS; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.05, Fisher Exact; Percentage Difference = 26.2 — For success rate with supplementation the difference between group US (98.2%) and group NS (72%) is 26.2%

ADVERSE EVENTS:
Arm/Group | Group US | Group NS
Serious Adverse Events (participants affected / at risk) | 0/125 | 1/125
Other Adverse Events (participants affected / at risk) | 66/125 | 24/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group US (N=125) | Group NS (N=125)
polyradicular sensomotor impairment (Nervous system disorders) | 0 (0) | 1 (1) — With one patient in the group NS, the insufficient block was supplemented by spinal anesthesia, which was initially free of complications. In the postoperative course polyradicular sensomotor impairment developed around lumbosacral plexus (L4-S1).
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group US (N=125) | Group NS (N=125)
Paresthesia (Nervous system disorders) | 66 (66) | 24 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No